CLINICAL TRIAL: NCT00289133
Title: Prospective, Comparative, Randomized Study of GVF Versus Cross-linked Polyethylene in Total Knee Arthroplasty
Brief Title: Gamma Vacuum Foil (GVF) Versus Cross-linked Polyethylene in Total Knee Arthroplasty Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03111
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis, Knee; Arthritis, Rheumatoid
Keywords: Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GVF (Active Comparator): Gamma Vacuum Foil polyethylene tibial insert
  Interventions: Device: total knee arthroplasty
- P.F.C. (Active Comparator): Cross-linked polyethylene tibial insert
  Interventions: Device: total knee arthroplasty

INTERVENTIONS:
Device: total knee arthroplasty — Gamma Vacuum Foil polyethylene tibial insert
  Arms: GVF
Device: total knee arthroplasty — cross-linked polyethylene tibial insert
  Other Names: P.F.C. Sigma cross-linked bearing
  Arms: P.F.C.

SUMMARY:
The purpose of this study is to evaluate long-term clinical and radiographic data between geometrically identical GVF and cross-linked polyethylene-bearing inserts in total knee arthroplasty.

DETAILED DESCRIPTION:
In 1996, Gamma Vacuum Foil (GVF) polyethylene was introduced as the first polyethylene to be gamma irradiated and packaged in an inert environment. This polyethylene, with its patented process and packaging, continues to be the only barrier-packaged process that is impermeable to both Hydrogen (H2) and Oxygen (O2), and allows the polyethylene to recombine and cross-link in the package. Though the new moderately cross-linked polyethylene being evaluated in this protocol is comparable to GVF geometrically and mechanically, the P.F.C.® Sigma™ cross-linked polyethylene also has the added benefit of being completely oxidatively stable both on the shelf and in-vivo.

The P.F.C. Sigma tibial tray component being assessed in this study is made of Cobalt Chrome (CoCr). The new CoCr tibial tray has the same design geometrically as the original titanium (Ti) tray, however, it features a highly polished top surface where it is joined to the polyethylene. This polished surface is designed to decrease the coefficient of friction between the polyethylene and the tray, thus minimizing backside wear. A comparative clinical study will be conducted to evaluate long-term clinical and radiographic data between geometrically identical cemented implants using GVF and crosslinked polyethylene tibial tray bearing inserts in Total Knee Arthroplasty (TKA) using the P.F.C. Sigma Total Knee System. Patients will be assigned to study treatment groups at random if they meet specific demographic and pathophysiologic criteria for cemented total knee arthroplasty. The anticipated duration of this investigation is a minimum six years, which includes a one-year enrollment phase.

The specific aims of this study are as follows:

1. Examine whether crosslinked polyethylene performs as well, if not better, than GVF polyethylene through standard clinical evaluations.
2. Evaluate long-term survivorship rates.
3. Report complications/adverse events.
4. Report radiographic findings of geometrically identical implants.

ELIGIBILITY:
Inclusion Criteria:

1. Osteoarthritis of the affected joint appropriate for Total Knee Arthroplasty.
2. Diagnosis of any of the following: rheumatoid or other inflammatory arthritis, post-traumatic arthritis, juvenile rheumatoid arthritis.
3. Radiographic evidence of sufficient sound bone stock to seat and support the prosthesis.
4. Subject requires a primary total knee replacement and is considered to be suitable for the specific knee prosthesis identified in protocol.
5. Subject has given consent to the transfer of his/her information to sponsor.
6. Subject will be compliant with requirements of protocol by returning for follow-up visits.

Exclusion Criteria:

1. History of recent/active joint sepsis.
2. Charcot neuropathy.
3. Psycho-social disorders that would limit rehabilitation.
4. Women who are pregnant or planning on being pregnant.
5. Greater than 80 years of age at the time of surgery.
6. Prior ipsilateral knee arthroplasty.
7. Metabolic disorders of calcified tissues, such as Paget's disease.
8. Severe diabetes mellitus that is not controlled by diet or oral agents.
9. Require joint replacement due to immunodeficiency syndromes.
10. Skeletal immaturity.
11. Avascular necrosis of the affected knee.
12. Chronic renal disease.
13. Subjects involved in medical-legal or worker's compensation claims.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 938 (Actual)
Dates: Start 2005-02-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gracia Etienne, MD, Principal Investigator — Orthopaedic & Spine Specialists; Michael L. Granberry, MD, Principal Investigator — Alabama Orthopaedic Clinic; Richard M. Konsens, MD, Principal Investigator — Jewett Orthopaedic Clinic
Locations (9):
- United States (9):
  - Alabama Orthopaedic Clinic, Mobile, Alabama
  - Pacific Bone and Joint Clinic, Berkley, California
  - Orthopedic Center of the Rockies, Fort Collins, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jewett Orthopaedic Clinic, Orlando, Florida
  - Jewett Orthopaedic Clinic, Winter Park, Florida
  - Loyola University, Chicago, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Orthopaedic & Spine Specialists, York, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- GVF Poly: Gamma Vacuum Foil polyethylene tibial component
- XLK Poly: Cross-linked polyethylene tibial component
Period: Overall Study
Arm/Group | GVF Poly | XLK Poly
Started | 461 | 477
Completed | 189 | 179
Not Completed | 272 | 298
Not completed — Non-study device implanted | 12 | 0
Not completed — Protocol Violation | 32 | 38
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Death | 5 | 10
Not completed — Lost to Follow-up - Hurricane Katri | 73 | 74
Not completed — Physician Decision | 41 | 45
Not completed — Revision | 8 | 6
Not completed — Lost to Follow-up | 92 | 115

BASELINE CHARACTERISTICS:
Population: Enrolled Subjects
Groups:
- GVF Poly: Gamma Vacuum Foil polyethylene tibial insert total knee arthroplasty: Gamma Vacuum Foil polyethylene tibial insert
- XLK Poly: Cross-linked polyethylene tibial insert total knee arthroplasty: cross-linked polyethylene tibial insert
- Total: Total of all reporting groups
Arm/Group | GVF Poly | XLK Poly | Total
Number analyzed (Participants) | 449 | 477 | 926
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (8.5) | 66.4 (8.5) | 66.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 290 | 308 | 598
  Male | 159 | 169 | 328
Region of Enrollment [Number; unit: participants]
  United States | 449 | 477 | 926

OUTCOME MEASURES:

1. Primary Outcome: Survivorship (Revision of Any Component for Any Reason)
Description: Survival was estimated by Kaplan-Meier method. Kaplan Meier survivorship analysis estimates the proportion of a population that will survive past a certain time avoiding a certain event. In this study, the event is removal of any component for any reason, also known as revision for any reason. Survival estimates are provided when 40 devices are left still being followed.
Time Frame: 5 years
Population: Survivorship can only be calculated on knees (not participants as some study subjects had bilateral knees in the study) with post-operative follow-up. 35 knees were excluded due to post-operative follow-up not being available. 67 knees were excluded due to protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of knees
Units Other Than Participants: number of knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 337 | 355
Number analyzed (number of knees) | 402 | 422
percentage of knees | 96.8 [93.9 to 98.4] | 98.1 [95.6 to 99.2]

2. Secondary Outcome: American Knee Society Evaluation - Total Score
Description: American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
Time Frame: 2 year
Population: The number of knees analyzed was the number available for analysis at this post-operative timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Knees
Groups:
- GVF Poly: Gamma Vacuum Foil polyethylene
- XLK Poly: Cross-linked polyethylene
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 240 | 239
Number analyzed (Knees) | 240 | 239
scores on a scale | 94.7 (7.9) | 93.5 (9.5)

3. Secondary Outcome: American Knee Society Evaluation - Total Score
Description: as for outcome 2
Time Frame: Minimum 5 years, up to 7.6 years
Population: The number of knees analyzed was the number available for analysis at this post-operative timepoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 145 | 146
Number analyzed (Knees) | 145 | 146
scores on a scale | 93.5 (9.2) | 93.1 (8.5)

4. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Osteoarthritis Total Score
Description: WOMAC is a patient reported outcome (PRO) that evaluates the condition of subjects with knee osteoarthritis, and includes pain (score range 0-20), stiffness (score range 0-8), and physical function (score range 0-68) of the joint. The total score ranged from 0 to 96. The subscales are combined (summed) to compute a total score, where a lower score indicates a better outcome.
Time Frame: 2 year
Population: The number of knees analyzed was the number available for analysis at this post-operative timepoint.
Measure: Mean (Standard Deviation); unit: scores (points) on a scale
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 225 | 221
Number analyzed (Knees) | 225 | 221
scores (points) on a scale | 10.2 (13.4) | 11.5 (15.3)

5. Secondary Outcome: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Osteoarthritis Total Score
Description: as for outcome 4
Time Frame: Minimum 5 years, up to 7.6 years
Population: The number of knees analyzed was the number available for analysis at this post-operative timepoint.
Measure: Mean (Standard Deviation); unit: scores (points) on a scale
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 139 | 134
Number analyzed (Knees) | 139 | 134
scores (points) on a scale | 11.0 (14.1) | 9.8 (13.2)

6. Secondary Outcome: Radiographic Outcomes - Percentage of Knees With Femoral Radiolucencies (>2mm)
Time Frame: Minimum 5 years, up to 7.6 years
Population: The number of knees analyzed was the number available for analysis at this post-operative timepoint.
Measure: Number; unit: percentage of knees
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 148 | 144
Number analyzed (Knees) | 148 | 144
percentage of knees | 9.5 | 7.6

7. Secondary Outcome: Radiographic Outcomes - Percentage of Knees With Tibial Radiolucencies (>2mm)
Time Frame: Minimum 5 years, up to 7.6 years
Population: The number of knees in which the radiographs were analyzed was the number available for analysis at this post-operative timepoint.
Measure: Number; unit: percentage of knees
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 148 | 144
Number analyzed (Knees) | 148 | 144
percentage of knees | 0 | 2.1

8. Secondary Outcome: Radiographic Outcomes - Percentage of Knees With Femoral Osteolysis (>2mm)
Time Frame: Minimum 5 years, up to 7.6 years
Population: The number of knees in which radiographs were analyzed was the number available for analysis at this post-operative timepoint.
Measure: Number; unit: percentage of knees
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 148 | 144
Number analyzed (Knees) | 148 | 144
percentage of knees | 0 | 0

9. Secondary Outcome: Radiographic Outcomes - Percentage of Knees With Tibial Osteolysis (>2mm)
Time Frame: Minimum 5 years, up to 7.6 years
Population: as for outcome 8
Measure: Number; unit: percentage of knees
Units Other Than Participants: Knees
Arm/Group | GVF Poly | XLK Poly
Number analyzed (Participants) | 148 | 144
Number analyzed (Knees) | 148 | 144
percentage of knees | 2.0 | 1.4

ADVERSE EVENTS:
Time Frame: Intraoperatively and postoperatively through 6 years.
Description: Since study inception, information on whether an adverse event (AE) was deemed to be serious was not collected. AE terms that are consistent with the definition of Serious AEs are included in the Serious AE table. Remaining AEs (serious or not) are included in the "Other" AE table. MedDRA was used to classify each AE into SOC, not Preferred Term.
Arm/Group | GVF Poly | XLK Poly
Serious Adverse Events (participants affected / at risk) | 16/461 | 15/477
Other Adverse Events (participants affected / at risk) | 146/461 | 164/477
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVF Poly (N=461) | XLK Poly (N=477)
Death (General disorders) | 5 (5) | 4 (4) — Unknown Cause
Death (Infections and infestations) | 2 (2) | 0 (0) — Complications from Septic Shock due to Necrotic Gallbladder and Bowel
Other - Had fall and fractured left shoulder and had a concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other - Flexion Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Revision of right total knee
Other - Left Hip Revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Underwent Total Hip Replacement after Breaking Hip
Other - Severe Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Led to Neurological Deficit
Other - Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Unknown Cause
Other - Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Other - Stage 4 Terminal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Other - Stage 4 Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Other - Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — From Respiratory Complications and Parkinson's Disease
Other - Death (Social circumstances) | 0 (0) | 1 (1) — Reported Suicide
Other - Follow-up Left Knee Arthroscope (Surgical and medical procedures) | 0 (0) | 1 (1)
Other - Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Other - Fall Injured Quad Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Dislocation (Product Issues) | 1 (1) | 2 (2)
Loosening (Product Issues) | 3 (3) | 0 (0)
Central Nervous System (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GVF Poly (N=461) | XLK Poly (N=477)
Cardiovascular (Cardiac disorders) | 7 (7) | 8 (9)
Other-Syncope Weakness (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 3 (3)
Musculoskeletal (General disorders) | 4 (17) | 4 (14)
Infection (Infections and infestations) | 6 (7) | 5 (5)
Central Nervous System (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal (Infections and infestations) | 0 (0) | 2 (3)
Other-Positive Nasal Culture for MRSA (Infections and infestations) | 1 (1) | 0 (0)
Wound Problem (Infections and infestations) | 3 (3) | 1 (1)
Musculoskeletal (Injury, poisoning and procedural complications) | 3 (4) | 5 (9)
Endocrine/Metabolic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Central Nervous System (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Endocrine/Metabolic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extensor Mechanism (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 30 (68) | 37 (87)
Other- Feeling of Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other-Follow-up right knee arthroscope (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other- Grade 1 Strain Medial Collateral Ligament (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other-Inflamed bursa over Gerdy's Tubercle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other-Mild Limp Secondary to Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other- Patella Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Other- Patella Clunk (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Other- Pes Bursitis; ITB syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other- Pesanserinus Tendonitis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Other- Pre Patellar Bursitis with Peri Patellar tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other- Routine F/U to Bilateral knee arthroscopic debulking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other- F/U Right Knee Arthroscope (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
other- Right Ankle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other- Subject has continuous right knee pain (non-surgical knee) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other- Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central Nervous System (Nervous system disorders) | 5 (6) | 7 (8)
Musculoskeletal (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Nervous System (Nervous system disorders) | 1 (1) | 1 (1)
Respiratory System (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Other- Dermis Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Other- Itchy Red Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other- Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other- Skin Rash on Low Bilateral Legs (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound Problem (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Other- Change in Insurance (Social circumstances) | 0 (0) | 1 (1)
Musculoskeletal (Surgical and medical procedures) | 10 (16) | 10 (12)
Peri-op AE - Other (Surgical and medical procedures) | 4 (4) | 8 (8)
Hematoma (Vascular disorders) | 2 (2) | 0 (0)
Pain (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis/Thrombophlebitis (Vascular disorders) | 6 (6) | 0 (0)
Stiffness, Arthrofibrosis, Ankylosis, Limited Range of Motion (Musculoskeletal and connective tissue disorders) | 12 (17) | 9 (9)
Other - Systemic: Voluntary Withdrawal (Social circumstances) | 0 (0) | 1 (2) — Reason not specified; Surgical Site not specified
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Endocrine/Metabolic (Endocrine disorders) | 0 (0) | 1 (1)
Central Nervous System (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 15 (19) | 17 (34)
Wound Problem (General disorders) | 0 (0) | 1 (1)
Gastrointestinal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hematological (Infections and infestations) | 1 (1) | 0 (0)
Hematological (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other - Advanced Alzheimer's (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Musculoskeletal (Product Issues) | 1 (2) | 1 (1)
Other - Radiographic subsidence of the femoral component - asymptomatic (Product Issues) | 1 (1) | 0 (0)
Genitourinary (Renal and urinary disorders) | 3 (3) | 3 (4)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Extensor Mechanism (Surgical and medical procedures) | 0 (0) | 1 (3)
Other - Left knee artrhoscopy (Surgical and medical procedures) | 0 (0) | 1 (2)
Musculoskeletal (Vascular disorders) | 0 (0) | 1 (1)
Other - Atraumatic onset of right buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Other - 20 degree flexion contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other - Bilateral knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Right knee pain greater than left knee pain; Arthroscope 2 months post-op
Other - Bilateral hand numbness and pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Carpal Tunnel Syndrome
Other - Fell and injured quad (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Serious adverse events were not collected in this study per the modern definition. All adverse events collected for this study will be reported in the 'Other Adverse Events' table. MedDRA was used to classify each AE into SOC, but not Preferred Term.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No